CLINICAL TRIAL: NCT05302960
Title: Recovering From COVID-19: Community-based Remote Monitoring in COVID-19 (SARS-CoV 2) Cases: The OVER-COVID Study
Brief Title: Recovering From COVID-19
Acronym: OVER-COVID
Status: Withdrawn | Type: Observational
Why Stopped: Decline in Covid Cases (not feasible to recruit)
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 21IC6755
Record Dates: First submitted 2022-03-29; First posted 2022-03-31 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: SARS CoV 2 Infection
Keywords: monitoring, ambulatory; vital signs; remote monitoring
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Fitbit — The use of Fitbit sensors to see if activity levels can be improved to track recovery from COVID

SUMMARY:
Following the success of pilot data trialling a virtual community-based remote monitoring model, using Bluetooth enabled pulse oximeters, which demonstrated a saving of 300 bed spaces over a three week period,9 a nationwide expansion is set to be implemented through NHS Digital. Participants who were on the virtual wards approximately 12 weeks after their admission and those referred to long-COVID outpatient clinics will be approached.

There is a particular lack of understanding as to whether post-COVID syndrome constitutes a singular disease process. It has been suggested that the post-COVID syndrome may be characterised into either an acute or chronic subtype, depending on whether symptoms extend beyond 12 weeks following initial diagnosis.7,10 However, it is not currently understood as to whether chronic post-COVID is either an extension of acute post-COVID or is a separate disease subtype that carries a distinct risk profile.

However, there remains a paucity in the literature depicting the recovery experience, risk factors for the development of post-COVID syndrome, management strategies, and qualitative experiences. This study aims to address these gaps

ELIGIBILITY:
INCLUSION CRITERIA

* Aged 18 years or over.
* Able to provide written consent.

EXCLUSION CRITERIA

* Any participants that withdraw their consent.
* Any form of psychiatric disorder or a condition that, in the opinion of the investigator, may hinder communication with the research team.
* Inability to cooperate or communicate with the research team.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: •Discharged from hospital with a RT-PCR SAR-CoV-2 positive swab result.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-11-30 (Estimated); Primary Completion 2024-04-08 (Estimated); Study Completion 2024-04-08 (Estimated)

PRIMARY OUTCOMES:
Step count | up to 1 year
  step count recorded from Fitbit devices